CLINICAL TRIAL: NCT02652936
Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Oral Doses of AF-130 in Healthy Subjects
Brief Title: A Pharmacokinetics Study of AF-130 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1112-001; AF130-001 (Other: Afferent)
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AF-130 capsule (Experimental): AF-130 oral capsules administered as a single dose or once daily for 7 days
  Interventions: Drug: AF-130
- AF-130 matching placebo capsule (Placebo Comparator): Oral placebo capsules to match AF-130 administered as a single dose or once daily for 7 days
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: AF-130 — AF-130 oral capsules (50 mg) administered as a single dose or once daily for 7 days
  Arms: AF-130 capsule
Drug: Placebo comparator — AF-130 matching placebo capsule
  Arms: AF-130 matching placebo capsule

SUMMARY:
This is a 2-part, single centre, single (Part 1) and multiple (Part 2) dose escalation study in healthy male subjects.

DETAILED DESCRIPTION:
Part 1 is a double-blind, placebo-controlled, randomised single dose design in up to 64 healthy male subjects. Part 1 will consist of Groups 1 to 6, each comprising 8 subjects (total of 48 subjects). There will be an option to enrol 2 additional groups (8 subjects in each of Groups 7 and 8) to assess alternative dose levels. Subjects will be randomised to receive active or placebo in the fasted state.

Part 2 is a double-blind, placebo-controlled, randomised, multiple ascending dose design in up to 45 healthy male subjects. Part 2 will consist of Groups 9 to 11, each comprising 9 subjects (total of 27 subjects). There will be an option to enrol 2 additional groups (9 subjects in each of Groups 12 and 13) to assess alternative multiple dose levels. Part 2 will not commence before completion of Groups 1 to 3 in Part 1. Subjects will be randomised to receive active or placebo in the fasted state. The planned dosing regimen is once per day however, this may be modified to twice per day depending on emerging pharmacokinetic data from Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age 18 to 55 years
* Body mass index of 18.0 to 35.0 kg/m2
* Willing and able to communicate and participate in the whole study
* Must provide written informed consent
* Must agree to use an adequate method of contraception

Exclusion Criteria:

* Participation in a clinical research study within the previous 3 months
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee
* Subjects who have previously been enrolled in this study
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
* Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening
* Subjects who do not have suitable veins for multiple venepunctures/cannulation
* Clinically significant abnormal biochemistry, haematology or urinalysis
* Positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* History of cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease as judged by the investigator
* QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 ms at screening and pre-dose
* Gastric or intestinal surgery, except for fully healed appendectomy and/or cholecystectomy
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment
* Ingestion of grapefruit or grapefruit juice within 48 h before dose administration
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol) or herbal remedies in the 14 days before study drug administration
* Receipt of an investigational product or device, or participation in a drug research study within a period of 30 days (or 5 half-lives, whichever is longer) before the first dose of study medication
* Receipt of an investigational immunomodulator or monoclonal antibody within 180 days (or 5 half-lives, whichever is longer) before the first dose of study medication
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-related adverse events following a single oral dose of AF-130 | 48 hours
Number of subjects with treatment-related adverse events following multiple oral doses of AF-130 | 7 days

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) profile of an oral formulation of AF-130 | 48 hours
Maximum plasma concentration (Cmax) profile of an oral formulation of AF-130 | multiple daily timepoints over 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Afferent Pharmaceuticals, Study Director — Afferent Pharmaceuticals Clinical Research
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom